CLINICAL TRIAL: NCT01578161
Title: The Effect of Dexmedetomidine on Emergence Agitation in Children Undergoing a Surgery Under Desflurane Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ah-Young Oh, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SNUBH_01
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Psychomotor Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dexmedetomidine0.25 (Experimental): dexmedetomidine 0.25 microg.kg(-1),(Group D0.25) ivs. for 10min.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine0.5 (Experimental): dexmedetomidine 0.5 microg.kg(-1),(group D0.5) ivs. for 10min.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine1.0 (Experimental): dexmedetomidine 1 microg.kg(-1) ivs. for 10min.
  Interventions: Drug: Dexmedetomidine
- NormalSaline (Placebo Comparator): Normal saline 10ml ivs. for 10min.
  Interventions: Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — There are four groups accoding to dosage of dexmedetomidine. Dexmedetomidine 0.25 microg.kg(-1),(group D0.25), dexmedetomidine 0.5 microg.kg(-1),(Group D0.5), dexmedetomidine 1 microg.kg(-1) (Group D 1) and normal saline(group P) is administered ivs. for 10mins when we are inducing each patient.
  Other Names: Precedex
  Arms: Dexmedetomidine0.25; Dexmedetomidine0.5; Dexmedetomidine1.0
Drug: 0.9% Normal Saline — Placebo,Normal saline 10ml ivs. for 10min.
  Arms: NormalSaline

SUMMARY:
After genernal anesthesia using sevoflurane or desflurane, the investigators can observe many cases of agiation (over 80%) and despite of no report of long-term complication, agitation is a big issue in PACU for doctors and nurses. The investigators use dexmedetomidine for prevention of agiation of preschool aged children. The investigators expect single injection of dexmedetomidine lead to decrease postoperative agitation and pain without any complication like oculocardiac reflex requiring atopine for treatment.

DETAILED DESCRIPTION:
There are four groups accoding to dosage of dexmedetomidine. Dexmedetomidine 0.25 microg.kg(-1),(group D0.25), dexmedetomidine 0.5 microg.kg(-1),(Group D0.5), dexmedetomidine 1 microg.kg(-1) (Group D 1) and normal saline(group P) is administered ivs. for 10mins when we are inducing each patient.

ELIGIBILITY:
Inclusion Criteria:

* Physical status classification of American Society of Anesthesiologist 1-2,
* Healthy, normal
* 2-6 years old
* Elective operation

Exclusion Criteria:

* Lack of consent
* Known adverse effects to dexmedetomidine, mental retardation
* Developmental delay, or neurological or psychiatric illness that may associate with agitation (cerebral palsy, seizure, etc)
* No cardiac disease

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Agitation score | 30 mins after operation

SECONDARY OUTCOMES:
Oculomotor reflex | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: AhYoung Oh, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, SEOUL NATIONAL UNIVERSITY BUNDANG HOSPITAL, SungNam-si, Kyonggi Do, South Korea